CLINICAL TRIAL: NCT05026060
Title: Measurement of Brain Perfusion by a Magnetic Resonance (MR) Perfusion Imaging Called eASL in Children's Cerebral Arteriopathies.
Brief Title: Measurement of Brain Perfusion by a MR Perfusion Imaging Called eASL in Children's Cerebral Arteriopathies.
Acronym: PEACE
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210339; 2021-A00225-36 (Other: IDRCB Number)
Record Dates: First submitted 2021-07-05; First posted 2021-08-30 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Arteriopathy
Keywords: Children's cerebral arteriopathies; Brain perfusion; Magnetic resonance (MR) perfusion imaging; ASL sequence with multiple post-labeling delays (eASL)
MeSH Terms: interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with arterial disease: Minor patients with acute or chronic arterial disease: diagnosis of Moyamoya, diagnosis of sickle cell disease, acute or chronic arterial infarction.
  Interventions: Diagnostic Test: Imaging

INTERVENTIONS:
Diagnostic Test: Imaging — 4-minutes eASL sequence without injection of contrast product added to each of the clinical MRs with standard ASL sequences performed for the care of the patient for 3 years.
  Other Names: eASL sequence

SUMMARY:
The MR sequence called MR-ASL is used to measure cerebral perfusion in children. This ASL sequence is used with a unique post-labeling delay (PLD) due to the technical impossibility of setting different post-labeling delays. The use of a single post-labeling, chosen by the pediatric radiology department of the Necker hospital, optimal in children without arteriopathy, may not be suitable for the lengthened arterial transit time of the spins marked in the pathological carotid network of a child with arterial disease.

Recently, ASL sequences with multiple delays (multi-PLD, called eASL) have been developed to overcome this limitation in arterial disease. To date, their use in the pre- and post-treatment evaluation of a child with acute or chronic arterial disease has not been evaluated.

The study hypothesis is that this eASL sequence is more efficient than single-delay ASL in measuring cerebral perfusion. The study will be performed in a population of children with acute or chronic arterial disease.

DETAILED DESCRIPTION:
For 9 years, the pediatric radiology department of the Necker Enfants Malades hospital has routinely used an MR sequence called MR-ASL, which has made it possible to measure cerebral perfusion in children. The service was a pioneer in using this sequence in children and it made it possible to detect areas of cerebral hypo-perfusion (or even pathological hyper-perfusion) and also to monitor post-surgical or spontaneous revascularizations. But this technique suffers from some limitations. Indeed, this ASL sequence is used with a unique post-labeling delay (PLD) of 1025 ms due to the technical impossibility of setting different post-labeling delays. This PLD corresponds to the arterial transit time of the spins marked to have a satisfactory cerebral perfusion. The use of a single post-labeling, chosen short (1025 ms) by the pediatric radiology department of the Necker hospital, optimal in children without arterial disease, may not be suitable for arterial transit time elongated spins marked in the pathological carotid network of a child with arterial disease.

Recently, ASL sequences with multiple delays (multi-PLD, called eASL) have been developed to overcome this limitation in arterial disease. To date, their use in the pre- and post-treatment evaluation of a child with acute or chronic arterial disease has not been evaluated.

The eASL is a sequence that lasts 4 minutes without injection of contrast product that the pediatric radiology department at Necker Hospital intends to add to the standard clinical sequences, as part of this study. This sequence will have no post-labeling delay a priori and will make it possible to test several post-labeling delays in one go. Thus, no a priori hypothesis on the transit time of the spins will be made and the eASL sequence will be able to show, after its reconstruction, what is the optimal post-labeling delay.

The study will be performed in a population of children with acute or chronic arterial disease. The study hypothesis is that this eASL sequence is more efficient than single-delay ASL in measuring cerebral perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Minor patients aged 0 to 18 with acute or chronic arterial disease: diagnosis of Moya-moya, diagnosis of sickle cell disease, acute and chronic arterial infarction.
* Necessity of diagnostic MR with standard ASL sequences for the care.
* Holders of parental authority and patients informed and not opposed to their participation in the study.

Exclusion Criteria:

* Usual contraindications to MR.
* Movement during ASL / eASL sequences.

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients with acute or chronic arterial disease followed at Necker hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Qualitative analysis of regional cerebral blood flow (CBF) in ASL and eASL based on a visual analysis of rainbow colored maps | 3 years
  In each parametric CBF map (ASL and eASL), brain regions appearing visually hypo- or hyperperfused compared to other brain regions will be recorded.
Quantitative analysis of regional cerebral blood flow (CBF) in ASL and eASL using Regions of Interest (ROIs) | 3 years
  In each parametric CBF map (ASL and eASL), the regional CBF will be measured in ml/100g/min over all brain regions by ROIs.
Quantitative analysis of regional cerebral blood flow (CBF) using statistical parametric map (SPM) | 3 years
  In each SPM processed CBF parametric map (ASL and eASL), regions with statistically significant hypo- or hyperflow compared to other regions will be recorded.

SECONDARY OUTCOMES:
Qualitative analysis of regional cerebral blood flow (CBF) change before and after surgical or spontaneous revascularization in ASL and eASL based on a visual analysis of rainbow colored maps | 3 years
  For each ASL sequence (ASL and eASL), pre-and post-revascularization parametric CBF maps will be displayed and co-registered. Brain regions visually showing variation in CBF after reperfusion compared with brain areas clear of acute or chronic arterial disease will be recorded.
Quantitative analysis of regional cerebral blood flow (CBF) variation before and after surgical or spontaneous revascularization in ASL and eASL using Regions of Interest (ROI) | 3 years
  For each ASL sequence (ASL and eASL), pre- and post-revascularization parametric CBF maps will be displayed and co-registered. In each brain region, the difference in CBF before and after revascularization (in ml/100g/min) will be measured using ROIs.
Quantitative analysis of regional cerebral blood flow (CBF) change before and after surgical or spontaneous revascularization in ASL and eASL unsing statistical parametric map (SPM) | 3 years
  Each ASL sequence (ASL and eASL) will be post-processed in SPM. Regions with a statistically significant change in CBF before and after revascularization will be recorded.
Optimal post-labeling delay | 3 years
  Calculation of optimal post-labeling delay (PLD) according to the type of arterial disease.
  Regional measures on the arterial transit time map.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie BODDAERT, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; David GREVENT, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No